CLINICAL TRIAL: NCT04069494
Title: Descriptors and Predictors of Burden and Information Needs on Symptom Self-management in Thai Patients With Lung Cancer and Their Family Caregivers During Palliative Radiotherapy
Brief Title: Descriptors and Predictors of Burden and Information Needs
Status: Completed | Type: Observational
Sponsor: Chulabhorn Cancer Center (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Saengrawee Thanthong, Principal Investigator, Chulabhorn Cancer Center
Other Study IDs: 200180015
Record Dates: First submitted 2019-08-02; First posted 2019-08-28 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Advanced Lung Cancer; Symptoms
Keywords: symptoms; predictor; information needs; self-management at home; palliative radiotherapy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: People diagnosed with advanced lung cancer and scheduled to receive palliative RT will be invited to participate between 1st July 2019 and 31st January 2020.
  Interventions: Other: questionnaires
- care giver: Patients' family caregivers will also be invited to participate
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Two questionnaires in patients and another two questionnaires in carer.

SUMMARY:
the purpose of this study is to investigate over time patients' symptom burden, caregiving burden, and patients and caregivers' need for information on patient symptom self-management at home during palliative radiotherapy(RT) for lung cancer. Repeatedly assessing burden and information needs on symptom self-management at home can help healthcare professionals to design a bespoke service and plan of care for both patients and family caregivers. In addition, I will explore psycho-social and clinical predictors of burden and information needs in patients and caregivers. These predictors can help health professionals to identify patients and caregivers at risk for distress during palliative radiotherapy for lung cancer.

DETAILED DESCRIPTION:
Eligible patients will be invited to take part in the study via a patient information sheet. They will also be asked to nominate their primary caregiver, who will also be invited to take part in the study. We will give patients and caregivers 24 hours to decide whether they want to take part or not. If they do decide to take part, all research participants will be involved in the study on four consecutive occasions before, during and after their treatment. These four time points will be the following:

* before first fraction of RT
* 1st week of RT (1st-5th faction)
* 2nd week of RT (6th-10th fraction)
* 1 month after the last fraction of RT The principal researcher, i.e. Saengrawee Thanthong, will endeavour to collect questionnaires in the hospital. If participants cannot come to the hospital to receive radiotherapy or for their follow up appointment and complete the questionnaire, then the principal researcher will call them and offer to complete the questionnaires over the phone so as to minimise missing data due to attrition.

ELIGIBILITY:
Inclusion Criteria:• Inclusion criteria for patients:

* Histological diagnosis of Lung cancer with stage III-IV(TNM)
* Age: 18 years or over
* Planning for palliative RT
* Scheduled to receive up to 10 fractions of palliative radiotherapy (Stevens, Macbeth, Toy, Coles, & Lester, 2015)

  • Exclusion criteria for patients:
* Non-English, Non-Thai speaking
* Diagnosis of severe cognitive or mental illness that affects communication

Patients' family caregivers will also be invited to participate as per below:

* Inclusion criteria for caregivers:

  * Family member of the care recipient can be spouse, child, parent, friend etc.
  * Age: 18 years or over
  * Only one family member if the patient presents with more than one.
  * Same person in every time point
* Exclusion criteria for caregivers:

  * Non-English, Non-Thai speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People diagnosed with advanced lung cancer and scheduled to receive palliative RT and their carer will be invited to participate between 1st september 2019 and 29 Febuary 2020.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Changes of symptom experiences | These four time points will be the following: before first fraction of RT, 1st week of RT (1st-5th faction), 2nd week of RT (6th-10th fraction) and 1 month after the last fraction of RT.
  Measure by the Thai version of modified version of the Memorial Symptom Assessment Scale (MSAS)
Changes of information need | These four time points will be the following: before first fraction of RT, 1st week of RT (1st-5th faction), 2nd week of RT (6th-10th fraction) and 1 month after the last fraction of RT.
  information need on symptom self-management at home measure by The Supportive Care Needs Survey - Patient version (SCNS) (Bonevski et al., 2000& McElduf et al., 2004) and Partners and Caregivers version (SCNS-P&C) - Information needs subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Saengrawee Thanthong, Principal Investigator — Mrs
Locations (1):
- ChulaBhorn Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bade BC, Thomas DD, Scott JB, Silvestri GA. Increasing physical activity and exercise in lung cancer: reviewing safety, benefits, and application. J Thorac Oncol. 2015 Jun;10(6):861-71. doi: 10.1097/JTO.0000000000000536. PMID 25831230
- [Background] Carnio S, Di Stefano RF, Novello S. Fatigue in lung cancer patients: symptom burden and management of challenges. Lung Cancer (Auckl). 2016 May 9;7:73-82. doi: 10.2147/LCTT.S85334. eCollection 2016. PMID 28210163
- [Background] Choi S, Ryu E. Effects of symptom clusters and depression on the quality of life in patients with advanced lung cancer. Eur J Cancer Care (Engl). 2018 Jan;27(1). doi: 10.1111/ecc.12508. Epub 2016 Apr 26. PMID 27112232
- [Background] Deshields TL, Potter P, Olsen S, Liu J. The persistence of symptom burden: symptom experience and quality of life of cancer patients across one year. Support Care Cancer. 2014 Apr;22(4):1089-96. doi: 10.1007/s00520-013-2049-3. Epub 2013 Dec 3. PMID 24292095
- [Background] Dionne-Odom JN, Hull JG, Martin MY, Lyons KD, Prescott AT, Tosteson T, Li Z, Akyar I, Raju D, Bakitas MA. Associations between advanced cancer patients' survival and family caregiver presence and burden. Cancer Med. 2016 May;5(5):853-62. doi: 10.1002/cam4.653. Epub 2016 Feb 10. PMID 26860217
- [Background] Kotronoulas G, Papadopoulou C, Burns-Cunningham K, Simpson M, Maguire R. A systematic review of the supportive care needs of people living with and beyond cancer of the colon and/or rectum. Eur J Oncol Nurs. 2017 Aug;29:60-70. doi: 10.1016/j.ejon.2017.05.004. Epub 2017 May 30. PMID 28720267
- [Background] Lee YH, Liao YC, Liao WY, Shun SC, Liu YC, Chan JC, Yu CJ, Yang PC, Lai YH. Anxiety, depression and related factors in family caregivers of newly diagnosed lung cancer patients before first treatment. Psychooncology. 2013 Nov;22(11):2617-23. doi: 10.1002/pon.3328. Epub 2013 Jul 28. PMID 23893960
- [Background] Lou VW, Chen EJ, Jian H, Zhou Z, Zhu J, Li G, He Y. Respiratory Symptoms, Sleep, and Quality of Life in Patients With Advanced Lung Cancer. J Pain Symptom Manage. 2017 Feb;53(2):250-256.e1. doi: 10.1016/j.jpainsymman.2016.09.006. Epub 2016 Nov 8. PMID 27832984
- [Background] Miaskowski C. Future Directions in Symptom Cluster Research. Semin Oncol Nurs. 2016 Nov;32(4):405-415. doi: 10.1016/j.soncn.2016.08.006. Epub 2016 Oct 21. PMID 27776833
- [Background] Morrison EJ, Novotny PJ, Sloan JA, Yang P, Patten CA, Ruddy KJ, Clark MM. Emotional Problems, Quality of Life, and Symptom Burden in Patients With Lung Cancer. Clin Lung Cancer. 2017 Sep;18(5):497-503. doi: 10.1016/j.cllc.2017.02.008. Epub 2017 Mar 2. PMID 28412094
- [Background] Rueda JR, Sola I, Pascual A, Subirana Casacuberta M. Non-invasive interventions for improving well-being and quality of life in patients with lung cancer. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD004282. doi: 10.1002/14651858.CD004282.pub3. PMID 21901689
- [Background] Schroder C, Engenhart-Cabillic R, Vorwerk H, Schmidt M, Huhnt W, Blank E, Sidow D, Buchali A. Patient's quality of life after high-dose radiation therapy for thoracic carcinomas : Changes over time and influence on clinical outcome. Strahlenther Onkol. 2017 Feb;193(2):132-140. doi: 10.1007/s00066-016-1068-7. Epub 2016 Oct 27. PMID 27787567
- [Background] Shallwani SM, Simmonds MJ, Kasymjanova G, Spahija J. Quality of life, symptom status and physical performance in patients with advanced non-small cell lung cancer undergoing chemotherapy: an exploratory analysis of secondary data. Lung Cancer. 2016 Sep;99:69-75. doi: 10.1016/j.lungcan.2016.06.018. Epub 2016 Jun 23. PMID 27565917
- [Background] Stapleton SJ, Holden J, Epstein J, Wilkie DJ. A Systematic Review of the Symptom Distress Scale in Advanced Cancer Studies. Cancer Nurs. 2016 Jul-Aug;39(4):E9-E23. doi: 10.1097/NCC.0000000000000292. PMID 26252436
- [Background] Sun V, Grant M, Koczywas M, Freeman B, Zachariah F, Fujinami R, Del Ferraro C, Uman G, Ferrell B. Effectiveness of an interdisciplinary palliative care intervention for family caregivers in lung cancer. Cancer. 2015 Oct 15;121(20):3737-45. doi: 10.1002/cncr.29567. Epub 2015 Jul 6. PMID 26150131
- [Background] Tan JY, Molassiotis A, Lloyd-Williams M, Yorke J. Burden, emotional distress and quality of life among informal caregivers of lung cancer patients: An exploratory study. Eur J Cancer Care (Engl). 2018 Jan;27(1). doi: 10.1111/ecc.12691. Epub 2017 Apr 18. PMID 28417550
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Wong ML, Cooper BA, Paul SM, Levine JD, Conley YP, Wright F, Hammer M, Miaskowski C. Differences in Symptom Clusters Identified Using Ratings of Symptom Occurrence vs. Severity in Lung Cancer Patients Receiving Chemotherapy. J Pain Symptom Manage. 2017 Aug;54(2):194-203. doi: 10.1016/j.jpainsymman.2017.04.005. Epub 2017 May 19. PMID 28533161
- [Background] Wong ML, Paul SM, Cooper BA, Dunn LB, Hammer MJ, Conley YP, Wright F, Levine JD, Walter LC, Cartwright F, Miaskowski C. Predictors of the multidimensional symptom experience of lung cancer patients receiving chemotherapy. Support Care Cancer. 2017 Jun;25(6):1931-1939. doi: 10.1007/s00520-017-3593-z. Epub 2017 Feb 3. PMID 28160076
- [Background] Yorke J, Lloyd-Williams M, Smith J, Blackhall F, Harle A, Warden J, Ellis J, Pilling M, Haines J, Luker K, Molassiotis A. Management of the respiratory distress symptom cluster in lung cancer: a randomised controlled feasibility trial. Support Care Cancer. 2015 Nov;23(11):3373-84. doi: 10.1007/s00520-015-2810-x. Epub 2015 Jun 26. PMID 26111954
- [Result] Chindaprasirt J, Limpawattana P, Pakkaratho P, Wirasorn K, Sookprasert A, Kongbunkiat K, Sawanyawisuth K. Burdens among caregivers of older adults with advanced cancer and risk factors. Asian Pac J Cancer Prev. 2014;15(4):1643-8. doi: 10.7314/apjcp.2014.15.4.1643. PMID 24641382
- [Result] Korner P, Ehrmann K, Hartmannsgruber J, Metz M, Steigerwald S, Flentje M, van Oorschot B. Patient-reported symptoms during radiotherapy : Clinically relevant symptom burden in patients treated with palliative and curative intent. Strahlenther Onkol. 2017 Jul;193(7):570-577. doi: 10.1007/s00066-017-1146-5. Epub 2017 Jun 1. PMID 28573475
- [Result] Mohile SG, Heckler C, Fan L, Mustian K, Jean-Pierre P, Usuki K, Sprod L, Janelsins M, Purnell J, Peppone L, Palesh O, Devine KA, Morrow G. Age-related Differences in Symptoms and Their Interference with Quality of Life in 903 Cancer Patients Undergoing Radiation Therapy. J Geriatr Oncol. 2011 Oct;2(4):225-232. doi: 10.1016/j.jgo.2011.08.002. PMID 22888384
- [Result] Reinke LF, Feemster LC, Backhus LM, Gylys-Colwell I, Au DH. Assessment and Management of Symptoms for Outpatients Newly Diagnosed With Lung Cancer. Am J Hosp Palliat Care. 2016 Mar;33(2):178-83. doi: 10.1177/1049909114557635. Epub 2014 Nov 5. PMID 25376224
- [Result] Zeng L, Koo K, Zhang L, Jon F, Dennis K, Holden L, Nguyen J, Tsao M, Barnes E, Danjoux C, Sahgal A, Chow E. Fatigue in advanced cancer patients attending an outpatient palliative radiotherapy clinic as screened by the Edmonton Symptom Assessment System. Support Care Cancer. 2012 May;20(5):1037-42. doi: 10.1007/s00520-011-1179-8. Epub 2011 May 4. PMID 21538097